CLINICAL TRIAL: NCT02079480
Title: Double-Blinded, Randomized, Placebo-Controlled, Single Ascending Dose and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986090 in Healthy Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, PK, and PD of BMS-986090 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IM142-003
Record Dates: First submitted 2014-03-04; First posted 2014-03-05 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — keyhole-limpet hemocyanin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Panel 1: BMS-986090 (0.5 mg) or Placebo (Experimental): BMS-986090 0.5 mg solution single dose subcutaneously once
  OR
  Placebo matching with BMS-986090 0 mg solution single dose subcutaneously once
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090
- Panel 2: BMS-986090 (3 mg) or Placebo (Experimental): BMS-986090 3 mg solution single dose subcutaneously once
  OR
  Placebo matching with BMS-986090 0 mg solution single dose subcutaneously once
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090
- Panel 3: BMS-986090 (10 mg) or Placebo (Experimental): BMS-986090 10 mg solution single dose subcutaneously once
  OR
  Placebo matching with BMS-986090 0 mg solution single dose subcutaneously once
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090
- Panel 4: BMS-986090 (30 mg) or Placebo + KLH (1 mg) (Experimental): BMS-986090 30 mg solution single dose subcutaneously once
  OR
  Placebo matching with BMS-986090 0 mg solution single dose subcutaneously once
  And Keyhole limpet hemocyanin (KLH) 1 mg solution single intramuscular dose once
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090; Drug: Keyhole limpet hemocyanin
- Panel 5: BMS-986090 (100 mg) or Placebo + KLH (1 mg) (Experimental): BMS-986090 100 mg solution single dose subcutaneously once
  OR
  Placebo matching with BMS-986090 0 mg solution single dose subcutaneously once
  And KLH 1 mg solution single intramuscular dose once
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090; Drug: Keyhole limpet hemocyanin
- Panel 6: BMS-986090 (100 mg) or Placebo (Experimental): BMS-986090 100 mg solution single dose intravenously once
  OR
  Placebo matching with BMS-986090 0 mg solution single dose intravenously once
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090
- Panel 7: BMS-986090 (300 mg) or Placebo + KLH (1 mg) (Experimental): BMS-986090 300 mg solution single dose subcutaneously once
  OR
  Placebo matching with BMS-986090 0 mg solution single dose subcutaneously once
  And KLH 1 mg solution single intramuscular dose once
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090; Drug: Keyhole limpet hemocyanin
- Panel 8: BMS-986090 (750 mg) or Placebo (Experimental): BMS-986090 750 mg solution single dose intravenously once
  OR
  Placebo matching with BMS-986090 0 mg solution single dose intravenously once
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090
- Panel 9: BMS-986090 (150 mg) or Placebo (Experimental): BMS-986090 150 mg solution subcutaneously once weekly for 4 weeks
  OR
  Placebo matching with BMS-986090 0 mg solution subcutaneously once weekly for 4 weeks
  Interventions: Drug: BMS-986090; Drug: Placebo matching with BMS-986090

INTERVENTIONS:
Drug: BMS-986090
Drug: Placebo matching with BMS-986090
Drug: Keyhole limpet hemocyanin
  Other Names: KLH
  Arms: Panel 4: BMS-986090 (30 mg) or Placebo + KLH (1 mg); Panel 5: BMS-986090 (100 mg) or Placebo + KLH (1 mg); Panel 7: BMS-986090 (300 mg) or Placebo + KLH (1 mg)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of BMS-986090 in healthy subjects.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Healthy male and female (of not childbearing potential), ages 18-45 years, inclusive
* BMI 18 to 32 kg/m2, inclusive

Exclusion Criteria:

- Any significant acute or chronic medical illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single dose measured by incidence, potential significance and clinical importance of AEs, as determined by medical review of AE reports, vital sign measurements, ECGs and results of physical examination and laboratory tests | Up to Day 85 after single dose of BMS-986090
  AE = Adverse event
  ECG = Electrocardiogram
Safety and tolerability of multiple dose measured by incidence, potential significance and clinical importance of AEs, as determined by medical review of AE reports, vital sign measurements, ECGs and results of physical examination and laboratory tests | Up to Day 106 after multiple dose of BMS-986090

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of BMS-986090 single dose subcutaneous (SC) and intravenous (IV) | Days 1 -85
Time of maximum observed serum concentration (Tmax) of single dose BMS-986090 SC and IV | Days 1 -85
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of single dose BMS-986090 SC and IV | Days 1 -85
Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of single dose BMS-986090 SC and IV | Days 1 -85
Terminal serum half-life (T-HALF) of single dose BMS-986090 SC and IV | Days 1 -85
Total body clearance (CLT) of single dose BMS-986090 IV | Days 1 -85
Apparent total body clearance (CLT/F) of single dose BMS-986090 SC | Days 1 -85
Volume of distribution at terminal phase (Vz) of single dose BMS-986090 IV | Days 1 -85
Volume of distribution during steady state (Vss) of single dose BMS-986090 IV | Days 1 -85
Apparent volume of distribution at terminal phase (Vz/F) of single dose BMS-986090 SC | Days 1 -85
Absolute bioavailability (F) of single dose BMS-986090 SC | Days 1 -85
Maximum observed serum concentration (Cmax) of multiple dose BMS-986090 SC | Days 1 -106
Time of maximum observed serum concentration (Tmax) of multiple dose BMS-986090 SC | Days 1 -106
Terminal serum half-life (T-HALF) of multiple dose BMS-986090 SC | Days 1 -106
Area under the serum concentration-time curve in one dosing Interval [AUC(TAU)] of multiple dose BMS-986090 SC | Days 1 -106
Trough observed plasma concentration (Ctrough) of multiple dose BMS-986090 SC | Days 1 -106
Average concentration over a dosing interval (Css-avg) of multiple dose BMS-986090 SC | Days 1 -106
Degree of Fluctuation (DF) of multiple dose BMS-986090 SC | Days 1 -106
AUC accumulation index (AI_AUC); ratio of AUC(TAU) at steady state to AUC(TAU) after the first dose of BMS-986090 SC (multiple dose) | Days 1 -106
Cmax accumulation index (AI_Cmax); ratio of Cmax at steady state to Cmax after the first dose of BMS-986090 SC (multiple dose) | Days 1 -106
Apparent total body clearance (CLT/F) of multiple dose BMS-986090 SC | Days 1 -106
Anti-KLH immunoglobulin G (IgG) and IgM antibody levels of single dose BMS-986090 SC | Days 1 -85
Immunogenicity of BMS-986090 following single SC / IV infusion measured by frequency of subjects with positive anti-drug-antibody (ADA) assessment and frequency of subjects who develop positive ADA following a negative baseline | Days 1 -85
Receptor occupancy (RO) of BMS-986090 following single SC or IV infusion | Days 1 -85

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - California Clinical Trials Medical Group, Glendale, California
  - Parexel Baltimore Early Phase Clinical Unit, Baltimore, Maryland

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx